CLINICAL TRIAL: NCT06690671
Title: An Open-Label, Single-Arm, Phase Ib Exploratory Study to Evaluate the Safety and Efficacy of Golidocitinib in Combination With Anti-PD-1 in Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) Treated With First-Line Anti-PD-1 Containing Regimens
Brief Title: A Single-Arm, Phase Ⅰb Study of Golidocitinib Combined With Anti-PD-1 for the Treatment of Previously Treated NSCLC
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Hua Zhong, Dr., Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS24147
Record Dates: First submitted 2024-11-14; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: JAKi; anti-PD-1; resitance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Golidocitinib in combination with anti-PD-1 (Experimental): Golidocitinib 150/75 mg once daily (QD) with anti-PD-1 （200 mg IV Q3W），21 days in one cycle.
  Interventions: Drug: Golidocitinib in combination with anti-PD-1

INTERVENTIONS:
Drug: Golidocitinib in combination with anti-PD-1 — Golidocitinib 150/75 mg once daily (QD) with anti-PD-1 （200 mg IV Q3W），21 days in one cycle.

SUMMARY:
This study is a phase Ib, single-center, single-arm exploratory clinical study designed to evaluate the safety and efficacy of Golidocitinib in combination with anti-PD-1 monoclonal antibody in locally advanced or metastatic NSCLC treated with anti-PD-1 in combination with or without platinum-containing chemotherapy regimens.

DETAILED DESCRIPTION:
This study is a phase Ib, single-center, single-arm exploratory clinical study designed to evaluate the safety and efficacy of Golidocitinib in combination with PD-1 monoclonal antibody in locally advanced or metastatic NSCLC treated with PD-1 monoclonal antibody in combination with or without platinum-containing chemotherapy regimens. The purpose of this part is to obtain the safety profile of the Golidocitinib in combination with PD-1 monoclonal antibody regimen in subjects with NSCLC who have failed treatment with first-line PD-1 monoclonal antibody in combination with or without platinum-containing chemotherapeutic regimens, and the recommended dose of the combination. The study will enroll 30 patients receiving Golidocitinib administered once daily (orally) at a starting dose of 75 mg up to a maximum dose of 150 mg; PD-1 monoclonal antibody at a clinically standardized dose (e.g., 200 mg IV Q3W), until the patients experienced disease progression, intolerable toxicity, or met the criteria for discontinuation of the trial drug. The primary endpoint was ORR, and secondary endpoints included PFS, DCR, OS, and safety. The study is expected to commence recruitment in mainland China in about Dec 2024. It is expected that the trial will end in July 2027.

ELIGIBILITY:
Inclusion Criteria:

1. be able to provide signed and dated informed consent, including adherence to the requirements and limitations listed in the Informed Consent Form (ICF) and in this protocol;
2. be ≥ 18 years of age, male or female, at the time of signing the ICF;
3. ECOG score of 0 or 1;
4. life expectancy ≥ 3 months;
5. patients with histologically or cytologically confirmed NSCLC diagnosed as locally advanced (Stage IIIB/IIIC), metastatic or recurrent (Stage IV) according to the International Association for the Study of Lung Cancer and the Joint Committee on the American Classification of Cancers, 8th edition of the TNM staging of lung cancer, who are not suitable for radical surgery or concurrent radiotherapy;
6. prior treatment with a first-line regimen of PD-1 monoclonal antibody (including, but not limited to, navulizumab, pabolizumab, treprostinil, sindilizumab, karelizumab, tirilizumab, and pegfilgrastimab) in combination with or without first-line regimen of platinum-containing chemotherapy, with a best-case outcome of CR/PR/SD that lasts at least 6 weeks;
7. intolerance to standard chemotherapy or refusal of chemotherapy;
8. at least one measurable lesion (RECIST v1.1);
9. adequate bone marrow reserve and organ system functional reserve, as summarized below:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L under conditions not receiving growth factor support.
   * Platelets ≥ 100 × 109/L under conditions of no growth factor support or transfusion.
   * Hemoglobin ≥ 9 g/dL without transfusion or receiving erythropoietin.
   * Total bilirubin ≤ 1.5 × ULN; if Gilbert syndrome (unconjugated hyperbilirubinemia) is present, total bilirubin should be ≤ 3 × ULN.
   * ALT and AST ≤ 2.5 × ULN; for patients with documented liver metastases, AST and ALT levels ≤ 5 × ULN.
   * Blood creatinine ≤ 1.5 × ULN, or creatinine clearance ≥ 50 mL/min calculated by the Cockcroft-Gault method, or urinary creatinine clearance ≥ 50 mL/min measured over 24 hours.
10. For patients with central nervous system metastases, the following conditions must be met for enrollment:

    * Absence of neurological symptoms or stabilization of symptoms for at least 2 weeks with local therapy, no need for corticosteroids or antiepileptic drugs, and cessation of hormone therapy within 3 days prior to the first study drug administration;
    * If the brain metastatic lesion has been treated locally (radiotherapy or surgery), there should be a window of ≥ 2 weeks prior to the first administration of study drug to ensure that adverse events related to local treatment have been reduced to CTCAE ≤ Grade 1.
11. Women of Childbearing Potential (WOCBP) must have a negative urine and/or serum (if the urine test is not confirmably negative) pregnancy test performed within 7 days prior to the first dose of study drug; the WOCBP or the man and his WOCBP partner should agree to take a urine and/or serum (if the urine test is not confirmably negative) pregnancy test from the time of signing the ICF until the last dose of 6 months after use of study drug to use effective contraception.

Exclusion Criteria:

1. histopathologically confirmed presence of a mixture of NSCLC and small cell lung cancer components;
2. the known presence of an EGFR-sensitive mutation/exon 20 insertion mutation or ALK/ROS1/RET fusion or MET14 jump mutation;
3. the known presence of interstitial pneumonitis/immune pneumonitis or interstitial changes
4. the known presence of spinal cord compression or meningeal metastases;
5. a history of any of the following:

   * Currently participating in an interventional clinical study treatment and any drug still in the developmental phase requiring a washout of 5 half-lives (or discuss with study team);
   * Received palliative radiotherapy within 2 weeks prior to the first dose, for more than 30% of the bone marrow for radiotherapy or extensive radiotherapy, which needs to be completed within 4 weeks prior to the first dose;
   * Currently receiving (or unable to discontinue use of) medications, herbal supplements, and foods known to be potent inducers or potent inhibitors of CYP3A at least 1 week prior to first dose;
   * Presence of an adverse event due to prior therapy via CTCAE > Grade 1 (with the exception of any degree of alopecia) prior to the first dose;
   * Known serious hematologic adverse event caused by a drug on prior first-line therapy that does not recover within 7 days to a Common Criteria for Terminology of Adverse Events (CTCAE) 5.0 rating of 2 or less.
6. receipt of a solid organ or hematologic transplant (e.g., previous allogeneic bone marrow transplant or whole blood transfusion within 120 days of sample collection during the study period)
7. subjects with severe pulmonary function decline (i.e., any FEV1 or DLCO < 60% of predicted). Prior interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis requiring steroid hormone therapy or current clinically active interstitial lung disease (including interstitial changes in the lungs), immunotherapy-induced immune pneumonitis of degree 3 or greater or resulting in treatment termination;
8. active autoimmune disease requiring systemic therapy (e.g., use of disease-mitigating drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency, etc.) are not considered systemic therapy;
9. physiologic doses of glucocorticoids (≤10 mg/day of prednisone or equivalent) are permitted for a diagnosis of immunodeficiency or if systemic glucocorticoid therapy or any other form of immunosuppressive therapy is being received within 7 days prior to the first dose of the study;
10. diagnosis of another malignancy within 5 years prior to the first dose, with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radically resected carcinoma in situ that has been evaluated and clinically cured;
11. vaccination with live vaccines, including live attenuated vaccines, except inactivated vaccines, within 30 days prior to the first dose (Cycle 1, Day 1);
12. active tuberculosis as determined by the Investigator, such as a positive tuberculin (PPD) test (nodule diameter > 10 mm), a positive T-SPOT test, a tuberculosis lesion on chest X-ray/CT, or other positive findings based on routine clinical screening (except for those cured by standardized anti-TB treatment as assessed by the Investigator);
13. subjects with active infections, including but not limited to hepatitis B virus (HBV), hepatitis C virus (HCV) human immunodeficiency virus (HIV); (1) Active HCV and HIV infection, i.e., positive test results for the respective antibodies; 2) Untreated active hepatitis B, defined as HBsAg-positive with HBV DNA ≥1000 IU/ml or HBcAb-positive with HBV DNA ≥1000 IU/ml; however, study participants who meet the following conditions may also be enrolled:

    * HBsAg-positive with HBV DNA <1000 IU/ml prior to the first dose of study drug, study participants should receive anti-HBV therapy to prevent viral reactivation throughout the study treatment period;
    * For HBsAg-negative, HBcAb-positive participants with HBV DNA <1000 IU/ml, study participants should be tested for HBV DNA throughout the duration of study treatment. 14.
14. hypersensitivity to the medications used in the study or their components;
15. have difficulty swallowing, or have an active digestive disorder, or have undergone major gastrointestinal surgery that may significantly interfere with the administration or absorption of the trial drug (e.g., ulcerative lesions, inability to swallow medications, uncontrollable nausea, vomiting, diarrhea, and malabsorption syndromes);
16. who, in the opinion of the investigator, are not suitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-15 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time from first dose to last dose, or up to 24 month
  To assess Golidocitinib overall response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as the proportion of subjects who have a complete response (CR) or a partial response (PR)

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from first subject dose to study completion, or up to 36 month
  To assess progression-free survival of patients treated by Golidocitinib according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator, define as first dose to first documented disease progression assessed by investigator or death due to any cause
Duration of Response (DoR) | Time from first subject dose to study completion, or up to 36 month
  To assess duration of response for subjects with CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 by investigator , defined as the time from the first documented CR or PR to disease progression or death
Overall survival (OS) | Time from first subject dose to study completion, or up to 36 month
  To assess overall survival, define as first dose to the death of the subject due to any cause
Adverse events (AEs) according to CTCAE 5.0 | From first dose until 28 days after the last dose, up to 24 month
  Number of participants with adverse events (AEs) according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- 241, West Huaihai Road, Shanghai, Shanghai, Shanghai 200030, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No